CLINICAL TRIAL: NCT03066349
Title: Conventional Ovarian Stimulation vs. in Vitro Oocyte Maturation (IVM) Followed by in Vitro Fertilisation (IVF): Differences in Patients' Emotional Adjustment and Quality of Life
Brief Title: IVM Versus IVF: Differences in Patients' Emotional Adjustment and Quality of Life
Acronym: EMAQOLIVMIVF
Status: Completed | Type: Observational
Sponsor: Universitair Ziekenhuis Brussel (Other)
Collaborators: University of the Basque Country (UPV/EHU) (Other)
Responsible Party: Principal Investigator, Michel De Vos, Kliniekhoofd en Klinisch Professor, Universitair Ziekenhuis Brussel
Other Study IDs: EMAQOL_2017
Record Dates: First submitted 2017-02-23; First posted 2017-02-28 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Infertility, Female; Polycystic Ovary Syndrome; Psychological Stress; Quality of Life
MeSH Terms: conditions — Infertility, Female; Polycystic Ovary Syndrome; Stress, Psychological | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with PCOS undergoing conventional ovarian stimulation
  Interventions: Other: Questionnaires
- Patients with PCOS undergoing IVM
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — FertiQoL and HADS (Hospital Anxiety and Depression Scale) questionnaires

SUMMARY:
Patients who undergo in vitro fertilization with or without intracytoplasmic sperm injection (IVF / ICSI) often experience an impact on their quality of life and emotional maladjustment to treatment and outcome. Multiple contributors to this negative impact have been identified, including interference with professional activities, expenses related to fertility treatment and hormonal side effects. In-vitro maturation (IVM) of human oocytes obtained from minimally stimulated or unstimulated ovaries offers a more "patient friendly" treatment option than the conventional ovarian stimulation protocols for Assisted Reproductive Technology (ART) treatment. Historically, IVM has been offered to women with increased ovarian response (so-called "high responders"), typically women with polycystic ovaries (PCO/PCOS), who are at increased risk for ovarian hyperstimulation syndrome (OHSS) if conventional ART protocols are used. IVM treatment programs are characterised by a minimal administration of fertility hormones, are less disruptive to patients' daily life through a reduced need for hormonal and ultrasound monitoring, avoid a range of minor and major complications because of the reduced hormonal burden of this procedure, and aim to reduce the total cost for of infertility treatment.

To facilitate the application of IVM as a treatment that can potentially improve the overall patient experience, a study comparing the psychological impact of a conventional ovarian stimulation protocol versus an IVM protocol will be conducted; furthermore, a study investigating the differences in quality of life between the two subgroups will also be performed.

Socio-demographic data, medical characteristics and the following questionnaires will be collected: Specific questions for patients with fertility problems (FertiQol); Hospital Anxiety and Depression Scale (HAD) and an instrument to measure side effects designed by the research group. The study group (IVF patients and IVM patients) will be evaluated at three predefined time points: at intake, after oocyte collection and when the outcome after the first embryo transfer is known.

Descriptive analysis, intergroup comparisons and explanatory/predictive model of the dependent variables (quality of life, emotional adjustment) will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Heterosexual or homosexual women enrolled to undergo ART treatment
* Patients with polycystic ovarian morphology (12 or more small follicles observed during a baseline pelvic ultrasound scan) or polycystic ovary syndrome (PCOS) (Rotterdam criteria, 2003)

Exclusion Criteria:

* Medical contra-indication for pregnancy
* High (>grade 2) grade endometriosis
* Patients who have previously undergone ART treatment
* Patients who require ART with PGD
* In vitro fertilisation with sperm retrieved through testicular biopsy
* Singles without a partner
* Couples who because of the language barrier (poor knowledge of Dutch, French or English) cannot reliably fill out the questionnaire.

Ages: 18 Years to 36 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Female infertility patients between 18 and 36 years.
Sampling Method: Non-Probability Sample
Enrollment: 149 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2023-04-06 (Actual); Study Completion 2023-04-06 (Actual)

PRIMARY OUTCOMES:
FertiQol score | 3 months
  Assessment of the influences of fertility problems in diverse life areas, for example, on general health, self-perceptions, emotions, partnership, family and social relationships, work life and future life plans.

SECONDARY OUTCOMES:
Hospital Anxiety and Depression Scale | 3 months
  Tool to determine the levels of anxiety and depression that a patient is experiencing

CONTACTS AND LOCATIONS:
Overall Officials: Michel De Vos, Principal Investigator — UZ Brussel - VUB
Locations (1):
- Universitair Ziekenhuis Brussel, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No